CLINICAL TRIAL: NCT02346565
Title: The Role of Contemporary Stress Echocardiography Techniques in the Initial Assessment of Women With No Previous History of Coronary Artery Disease (CAD) Who Present With Chest Pain of Recent Onset. Stress Echocardiography vs Exercise ECG as First Line Investigation in This Population. Potential for Higher Diagnostic Accuracy Cost Saving.
Brief Title: Stress Echocardiography Versus Exercise ECG (ExECG) in Women With Chest Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RD14/86
Record Dates: First submitted 2015-01-14; First posted 2015-01-27 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise ECG (Other): Patients will undergo an exercise test using the standard Bruce protocol. Standard end points of exercise testing will include: fatigue, severe ischaemia (severe chest pain, >2mm ST depression on ECG), hypertension (systolic BP>220mmHg), hypotension, pre-syncope or arrhythmia.
  Interventions: Procedure: Exercise ECG
- Stress Echocardiography (Other): A two-dimensional echocardiogram will be performed in the lateral decubitus position. Digitized images of the left ventricle (LV) will be obtained in the parasternal long-axis, short-axis, and apical four-, two-, and three-chamber views.
  In the case of exercise stress echo, images will be acquired at rest and immediately (within 90 seconds) after peak exercise.
  In the case of dobutamine stress echo, images will be acquired at rest, at the end of stage one of dobutamine administration (10mcg/Kg/min) and at peak stress.
  Interventions: Procedure: Stress Echocardiography

INTERVENTIONS:
Procedure: Exercise ECG
  Arms: Exercise ECG
Procedure: Stress Echocardiography
  Arms: Stress Echocardiography

SUMMARY:
The overall question the investigators would like to help answer is whether SE with or without MCE data can be widely used as a first line investigation in women with no previous history of Coronary Artery Disease (CAD) who present with chest pain of recent onset. In order to answer this question the investigators will look at the following:

i) Is SE superior to ExECG in terms of cost to diagnosis and negative predictive value of CAD?

ii) What is the additive value of myocardial perfusion data to wall motion data for predicting significant CAD on angiography and future cardiac events in women?

iii) What is the additive value of Carotid ultrasonography in a large population of women referred for stress testing?

DETAILED DESCRIPTION:
The investigators plan to perform a prospective study on all women seen in our RACPC with no previous history of CAD and intermediate pre-test probability of CAD as determined by National Institute for Health and Care Excellence (NICE) guidelines, who require a functional test as part of their assessment. All patients that meet the inclusion criteria and do not meet any of the exclusion criteria will be approached for consent to the study.

Patients who can perform greater than 5 metabolic equivalents (METS) on the Duke Activity Status Index (DASI) questionaire will be randomised between undergoing an Exercise ECG (Ex-ECG) or Exercise Stress Echo (ESE). The DASI is a 12-item questionnaire that estimates self-reported physical work capacity and is converted to an estimate of peak metabolic equivalents. Patients who do not meet this criteria, will undergo a pharmacological stress echocardiogram using Dobutamine (DSE), including Myocardial Contrast Echocardiography (MCE). Investigations will continue to be performed as per standard clinical departmental protocols as described below. In addition, all patients will undergo carotid ultrasonography. The techniques used are described for completeness as they are all well-established in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 years and above
* No previous history of Coronary Artery Disease
* Chest pain of presumed cardiac origin, which has occurred in the last month prior to the clinic appointment.

Exclusion Criteria:

* Electrocardiogram diagnostic of cardiac ischaemia and/or infarction (ST-segment deviations>0.5mm, or T-wave inversion).
* Previous history of Coronary Artery Disease
* Chest pain in the last 24 hours
* Inability to provide informed consent
* Pregnancy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2015-01; Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
Comparison of Positive Predictive Value of each test for Coronary artery disease detection | 2 years
  To compare positive predictive value of each test for the detection of obstructive CAD defined as ≥ 70% luminal diameter narrowing in one or more epicardial coronary arteries or their major branches during invasive coronary arteriography
To compare the use of Downstream resource utilisation following allocated functional tests | 2 years
  Comparison between the number of follow-up investigations, clinic visits and hospitalisation for patients in the 2 test groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwick Park Hospital, Harrow, Middx, United Kingdom